CLINICAL TRIAL: NCT05691946
Title: Acute Effects of Kinesiology Taping On Functional Performance And Physical Parameters In Handball Players: Randomised Placebo-Controlled Trial
Brief Title: Acute Effects of Kinesiology Taping in Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: AmasyaU12
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Kinesiology Taping
Keywords: muscle strength; proprioception; handball players

STUDY DESIGN:
Intervention Model Description: A randomised placebo-controlled with pretest-posttest both groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: It was a double blinded study:
  * Participants were blind to the taping (sham taping or kinesiology taping).
  * Outcome assessor was blind to the participants' group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology Taping Group (Experimental): Kinesiology Taping Group
  Interventions: Procedure: Kinesiology Taping
- Placebo Control Group (Placebo Comparator): Placebo Taping Group
  Interventions: Procedure: Placebo Taping

INTERVENTIONS:
Procedure: Kinesiology Taping — The experimental group was applied 'Y shaped' kinesiology taping on gastro-soleus muscle group, based on facilitation technique with 25-50% stretching.
  Arms: Kinesiology Taping Group
Procedure: Placebo Taping — The placebo group was applied kinesiology taping on gastro-soleus muscle group without any stretching.
  Arms: Placebo Control Group

SUMMARY:
The aim of this randomised placebo-controlled study was to investigate the acute effect of kinesiology taping in the gastro-soleus muscle group of handball players.

Researchers compared the placebo and the kinesiology taping groups to see if there were any effects on foot plantar and dorsiflexion muscle strength, balance, proprioception, horizontal jumping and injury proneness.

DETAILED DESCRIPTION:
This randomised placebo-controlled and double blinded study aimed to investigate the acute effect of kinesiology taping in the gastro-soleus muscle group, which has the key role in jumping, of handball players on foot plantar and dorsiflexion muscle strength, balance, proprioception, horizontal jumping and injury proneness. There were two groups in the study: the experimental group was applied 'Y shaped' kinesiology taping on gastro-soleus muscle group, based on facilitation technique with 25-50% stretching. The control (placebo) group was applied kinesiology taping on gastro-soleus muscle group without any stretching. Participants' muscle strength, proprioception, balance, horizontal jumping and injury proneness was measured before and two hours after taping.

ELIGIBILITY:
Inclusion Criteria:

* Licensed handball player
* Volunteer to participate the study

Exclusion Criteria:

* Any discomfort that is contraindicated for the measurements
* Have suffered any injury in the last 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 2 hours
  Foot dorsiflexion and plantar flexion muscle strength were measured using a manual dynamometer (MicroFET2 (Hogan Inc., West Jordan, USA). This device; shows the peak force in Newtons on its own screen. Measurements were made in three repetitions after a 30-second records. The highest value was recorded.
Proprioception | 2 hours
  Ankle proprioception was measured using Baseline Digital Inclinometer (New York, USA) device. This was measured on the dominant and non-dominant ankle with eyes open and eyes closed. Ankle dorsiflexion at 10 degrees, ankle plantar flexion at 11 degrees, and 25 degrees was measured in active reproduction test positions.

SECONDARY OUTCOMES:
Horizontal jump performance | 2 hours
  This was measured by standing long jump with the direction of movement develops from vertical to horizontal. The distance between the zero point and the last point of contact of the foot was measured in centimetres. Three repetitions were performed and the highest value was recorded.
Balance | 2 hours
  Dynamic balance was measured with Y-balance test. The participant reached anterior, posteromedial, and posterolateral directions with one foot, while other foot was on the centre. The test was repeated three times in each direction and the average was recorded in centimetres.
Injury proneness | 2 hours
  Injury proneness was measured using Functional Movement Screen test. This test consists of seven different positions to measure strength, flexibility, balance and such various motor skills. The movements are deep squats, high stepping, single-line stepping forward, shoulder mobility, active straight leg raise, trunk stability push-ups, rotation stability. Each movement is scored between 0 and 3 points, the score that the participant can get from the test is between 0 and 21. It was scored 3 points if the movement was performed completely well, 2 points if the movement was performed with an error, 1 point if the movement was not performed according to the specified instruction, and 0 points if pain was experienced during the movements.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No